CLINICAL TRIAL: NCT03448315
Title: Role of Transcrainal Direct Current Brain Stimulation in Acute and Chronic Post-mastectomy Pain Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shereen Mamdouh, Lectruer of anesthesia, ICU and pain manegement, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 405
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Postoperative Pain
Keywords: brain stimulation, tDCS, acute postoperative pain, chronic pain
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real tDCS (Active Comparator): motor cortex stimulation (2 mA, 20 min for 4 sessions)
  Interventions: Device: tDCS
- sham tDCS (Sham Comparator): motor cortex stimulation (2 mA, 20 min for 4 sessions) but stimulation device is turned off without the participant knowledge
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — motor cortex stimulation (2 mA, 20 min for 4 sessions)

SUMMARY:
the role of transcranial magnetic stimulation over the primary motor cortex area on acute postoperative pain after breast cancer surgery and on the probability of developing chronic neuropathic pain.

DETAILED DESCRIPTION:
New analgesic strategies are needed that can be used adjunctively to existing strategies with the potential to reduce reliance on opioid analgesia. Several novel brain stimulation technologies including transcranial direct current stimulation (tDCS) are beginning to demonstrate promise as treatments for a variety of pain conditions. Electricity has no metabolite or other residue, and can be delivered with minimal discomfort and without problems associated with drug-drug interactions.Transcranial direct current stimulation has been studied in patients with various disorders and multiple pain syndromes. There is also evidence that tDCS might be useful in postsurgical pain reduction.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II, scheduled for unilateral modified radical mastectomy with axillary dissection for breast cancer

Exclusion Criteria:

* patients with intracranial metallic devices or with pacemakers or any other device.
* patients with Neurological or psychiatric disorders,
* patients taking major centrally acting drugs (antiepileptics or antidepressants), -opioid dependence,
* substance abuse,
* severe cardiopulmonary, renal, hepatic diseases, and
* those with extensive myocardial ischemia or unstable angina.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-12-02 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
total morphine comsuption | 48 hours
  the total dose of morphine used as analgesic expressed in mg

SECONDARY OUTCOMES:
Visual analogue scale | baseline,at 2,4,6, 12, 24,36,48 hours
  patient asked to describe this pain with scores ranging from 0 to10 (with 0 = no pain and 10 = the worst pain imaginable)
Douleur Neuropathique 4 questions DN4 | 1month, 3month, 6 month
  the possibility of development of neuropathic pain will be assessed using DN4 scale

CONTACTS AND LOCATIONS:
Locations (1):
- South Egypt Cancer Institute, Asyut, Egypt